CLINICAL TRIAL: NCT02151760
Title: Study of 18F-DCFPyL, a Second Generation Low-molecular Weight PSMA-based PET Radiotracer, in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1418; NA_00092956 (Other: JHMIRB); P50CA103175 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

ARMS (1):
- 18F-DCFPyL (Experimental)
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL
  Other Names: 10.0 A bolus of less than or equal to 9 mCi (331 MBq) of 18F-DCFPyL will be injected into the IV line by slow push IV push.

SUMMARY:
This study is being done to determine the safety, biodistribution, and radiation dosimetry of 18F-DCFPyL, and to detect prostate cancer by visual analysis.

DETAILED DESCRIPTION:
To assess the hypothesis that this new 2nd generation positron emission tomography (PET) radiopharmaceutical, 18F-DCFPyL, may possess pharmacokinetic and pharmacodynamic properties that will represent an advance in imaging metastatic prostate cancer in ten patients diagnosed with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be enrolled into this protocol only if all of the following inclusion criteria are met:

  1. Greater than or equal to 18 years of age
  2. Histological confirmation of prostate cancer
  3. Radiologic evidence of new or progressive metastatic disease demonstrated on anatomical imaging (CT, MRI, or ultrasound), bone scintigraphy, 18F-Sodium Fluoride PET, or 18F-FDG PET
  4. PSA ≥ 1.0 ng/mL
  5. Can be on androgen deprivation therapy if dose is stable for ≥ 1 week.
  6. Platelet count > 50,000/mm3
  7. Neutrophil count > 1,000/mm3
  8. Patient is judged by the Investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits.
  9. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures.

Exclusion Criteria:

* Patients will be excluded from enrollment if any of the following apply:

  1. Karnovsky performance status of < 60
  2. Inadequate venous access (two antecubital or equivalent venous access sites are required for study drug injection and PK blood sampling, respectively)
  3. Patient received a permanent prostate brachytherapy implant within the last 3 months (for Pd-103 implants) or 12 months (for I-125 implants)
  4. Administered a radioisotope within 5 physical half-lives prior to study enrollment
  5. Serum creatinine > 3 times the upper limit of normal
  6. Total bilirubin > 3 times the upper limit of normal
  7. Liver Transaminases > 5times the upper limit of normal
  8. Patient has been treated with an investigational drug, investigational biologic, or investigational therapeutic device within 30 days prior to study radiotracer administration
  9. Prior radiation therapy or chemotherapy within 2 weeks prior to study radiotracer administration (Washout is one half-life of the drug or 2 weeks, whichever is longest).
  10. Prior history of any other malignancy within 3 years, other than skin basal cell carcinoma.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
PET/CT Detection of Metastatic Disease | 12 months
  To comare diagnostic accuracy of 18-DCFPyL to CIM(CT and bone scintigraphy) for the detection of metastatic prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Y Cho, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States